CLINICAL TRIAL: NCT01691482
Title: A 4-Week Randomized Cross-Over Study to Evaluate Daily Lung Function Following the Administration of Albuterol/Salbutamol and Ipratropium in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Look at Day to Day Changes in Lung Function in COPD Subjects Taking Albuterol/Salbutamol and Ipratropium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 114956
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Ipratropium

ARMS (2):
- Albuterol/salbutamol followed by ipratropium (Active Comparator): Subjects will recieve daily albuterol/salbutamol followed by ipratropium which will be adminstered one hour after adminstration of albuterol/salbutamol
  Interventions: Drug: Albuterol/salbutamol
- Ipratropium followed by albuterol/salbutamol (Active Comparator): Subjects will recieve daily ipratropium followed by albuterol/salbutamol which will be adminstered one hour after adminstration of ipratropium
  Interventions: Drug: Ipratropium

INTERVENTIONS:
Drug: Albuterol/salbutamol — Albuterol/salbutamol (daily)
  Arms: Albuterol/salbutamol followed by ipratropium
Drug: Ipratropium — Ipratropium (daily)
  Arms: Ipratropium followed by albuterol/salbutamol

SUMMARY:
The objective of this study is to assess the daily variation in bronchodilator response to an inhaled short acting beta2-agonist (albuterol/salbutamol) and an inhaled short acting anticholinergic (ipratropium) individually and when used in combination in subjects with COPD.

DETAILED DESCRIPTION:
Beta2-agonist and anticholinergics are a principle component of the pharmacologic management of chronic obstructive pulmonary disease COPD. It has been demonstrated that the combination of a short acting beta2-agonist and a short acting anticholinergic yields greater efficacy as measured by FEV1 when compared with the response to the individual short acting bronchodilators. However, daily bronchial response to these agents is poorly understood. It is also poorly understood how the variation in magnitude of the response to the individual agents and how the variation in response for one agent coincides with the variation in response to the other agent. This study will seek to define the pattern of response of each individual agent and the relationship between them. The study will also explore if the combination of the two agents leads to less variation in response compared to the individual agents. This is a randomized, open label, two period cross-over study. Eligible subjects will be randomized to a sequence of either albuterol/salbutamol via metered-dose inhaler (MDI) followed by ipratropium via MDI or the same dose of each bronchodilator given in the opposite order. Each study period will consist of 10 clinic visits to be conducted over 10 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give their signed and dated written informed consent to participate.
* Subjects 40 years of age or older at Visit 1.
* Male or female subjects .
* An established clinical history of COPD.
* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at Visit 1.
* A post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and a post-albuterol/salbutamol FEV1 of >=30 and <= 70% of predicted normal values at Visit 1 calculated using NHANES III reference equations .

Exclusion Criteria:

* A current diagnosis of asthma
* Women who are pregnant of lactating or are planning on becoming pregnant during the study.
* Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Participation in pulmonary rehabilitation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-07-23; Primary Completion 2012-10-01 (Actual); Study Completion 2012-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Spartanburg, South Carolina, United States
- GSK Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Singh D, Zhu CQ, Sharma S, Church A, Kalberg CJ. Daily variation in lung function in COPD patients with combined albuterol and ipratropium: results from a 4-week, randomized, crossover study. Pulm Pharmacol Ther. 2015 Apr;31:85-91. doi: 10.1016/j.pupt.2014.08.010. Epub 2014 Sep 6. PMID 25197005
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomized, open-label, two-period cross-over study to evaluate the daily bronchodilator response to albuterol/salbutamol and ipratropium individually and in combination in participants with chronic obstructive pulmonary disease.
Groups:
- A/S Then Ipratropium in TP1; Ipratropium Then A/S in TP2: Participants received albuterol (4 puffs; 90 micrograms [µg] per puff)/salbutamol (A/S) (4 puffs; 100 µg per puff) followed by ipratropium (4 puffs; 20 µg per puff) via a metered-dose inhaler (MDI) during treatment period 1 (TP1) then, ipratropium followed by A/S at the same doses via an MDI in treatment period 2 (TP2).
- Ipratropium Then A/S in TP1; A/S Then Ipratropium in TP2: Participants received Ipratropium (4 puffs; 20 µg per puff) followed by albuterol (4 puffs; 90 µg per puff)/salbutamol (4 puffs; 100 µg per puff) (A/S) via a MDI in TP1, then A/S followed by ipratropium at the same doses via an MDI in TP2.
Period: Treatment Period 1
Arm/Group | A/S Then Ipratropium in TP1; Ipratropium Then A/S in TP2 | Ipratropium Then A/S in TP1; A/S Then Ipratropium in TP2
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | A/S Then Ipratropium in TP1; Ipratropium Then A/S in TP2 | Ipratropium Then A/S in TP1; A/S Then Ipratropium in TP2
Started | 28 | 28
Completed | 27 | 26
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All participants randomized to receive a sequence of either salbutamol (4 puffs; 100 µg per puff) via an MDI and albuterol (4 puffs; 90 µg per puff) followed by ipratropium (4 puffs; 20 µg per puff) via an MDI in TP1 and the same dose of each bronchodilator given in the opposite order in TP2, or ipratropium followed by albuterol/salbutamol in TP1 and the same dose of each bronchodilator given in the opposite order in TP2
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 4
  White | 52

OUTCOME MEASURES:

1. Primary Outcome: Variability in Daily FEV1, Estimated by Coefficient of Variation
Description: FEV1 is the maximal amount of air that can be forcefully exhaled in one second. During each study period, pre- and post-bronchodilator spirometry for evaluation of FEV1 was performed at study visits as follows: prior to administration of the first short-acting bronchodilator, approximately 1 hour after administration of the first bronchodilator (1 hour), and approximately 1 hour after administration of the second short-acting bronchodilator (2 hours). Variability in daily FEV1 was measured as the fluctuation around the mean FEV1 data collected from Day 1 to Day 10. Variability was measured by the coefficient of variation (CV) and the half range. The CV is the dispersion of the data around the mean, whereas the half range method is the difference between the maximum and minimum FEV1 values.
Time Frame: up to 10 days
Population: Efficacy Population: participants in the Intent-to-Treat Population (all participants who were randomized and received at least one bronchodilator in the treatment period) who completed pre- and post- bronchodilator assessments for at least 17 visits, with no more than 3 consecutive missing days
Measure: Mean (Standard Error); unit: Liters
Groups:
- Albuterol/Salbutamol Followed by Ipratropium: All participants randomized to receive a sequence of albuterol (4 puffs; 90 µg per puff)/salbutamol (4 puffs; 100 µg per puff) via an MDI followed by ipratropium (4 puffs; 20 µg per puff) via an MDI in either TP1 or TP2.
- Ipratropium Followed by Albuterol/Salbutamol: All participants randomized to receive a sequence of ipratropium (4 puffs; 20 µg per puff) via an MDI followed by albuterol (4 puffs; 90 µg per puff)/salbutamol (4 puffs; 100 µg per puff) via an MDI in either TP1 or TP2
Arm/Group | Albuterol/Salbutamol Followed by Ipratropium | Ipratropium Followed by Albuterol/Salbutamol
Number analyzed (Participants) | 55 | 55
Liters
  Pre-dose/non-bronchodilator | 0.081 (0.0394) | 0.079 (0.0372)
  Albuterol/Salbutamol (A/S) alone, 1 hour | 0.059 (0.0276) | NA (NA) — Participants in this treatment arm received ipratropium as the first bronchodilator; thus, data were not collected for albuterol/salbutamol (A/S) at this time point.
  A/S followed by ipratropium, 2 hours | 0.054 (0.0232) | NA (NA) — Participants in this treatment arm received ipratropium followed by A/S; thus, data were not collected for A/S followed by ipratropium.
  Ipratropium alone, 1 hour | NA (NA) — Participants in this treatment arm received A/S as the first bronchodilator; thus, data were not collected for ipratropium at this time point. | 0.072 (0.0406)
  Ipratropium followed by A/S, 2 hours | NA (NA) — Participants in this treatment arm received A/S followed by ipratropium; thus, data were not collected for ipratropium followed by A/S. | 0.063 (0.0327)
Statistical Analysis 1: Comparison: Albuterol/Salbutamol Followed by Ipratropium; Test type: Superiority or Other; Adjusted Mean = 0.058, 95% CI [0.049 to 0.067], Standard Error of Mean 0.0046 — Treatment: A/S alone. A mixed model analysis, with period, treatment (A+I, I+A, Albuterol alone, Ipratropium alone), FEV1 Baseline, smoking status at Screening, and center fitted as fixed effects and participant as a random effect was used
Statistical Analysis 2: Comparison: Ipratropium Followed by Albuterol/Salbutamol; Test type: Superiority or Other; Adjusted Mean = 0.071, 95% CI [0.062 to 0.080], Standard Error of Mean 0.0046 — Treatment: ipratropium alone. A mixed model analysis, with period, treatment (A+I, I+A, Albuterol alone, Ipratropium alone), FEV1 Baseline, smoking status at Screening, and center fitted as fixed effects and participant as a random effect was used
Statistical Analysis 3: Comparison: Albuterol/Salbutamol Followed by Ipratropium; Test type: Superiority or Other; Adjusted Mean = 0.053, 95% CI [0.044 to 0.062], Standard Error of Mean 0.0046 — Treatment: A+I. A mixed model analysis, with period, treatment (A+I, I+A, Albuterol alone, Ipratropium alone), FEV1 Baseline, smoking status at Screening, and center fitted as fixed effects and participant as a random effect was used
Statistical Analysis 4: Comparison: Ipratropium Followed by Albuterol/Salbutamol; Test type: Superiority or Other; Slope = 0.062, 95% CI [0.053 to 0.071], Standard Error of Mean 0.0046 — Treatment: I+A. A mixed model analysis, with period, treatment (A+I, I+A, Albuterol alone, Ipratropium alone), FEV1 Baseline, smoking status at Screening, and center fitted as fixed effects and participant as a random effect was used

2. Secondary Outcome: The Maximal Bronchodilator Response for the First Administered Agent
Description: The maximal bronchodilator response for the first administered agent is defined as the FEV1 (the maximal amount of air that can be forcefully exhaled in one second) 1 hour post-dose of the first bronchodilator minus the pre-dose. The maximal bronchodilator response for the second agent is defined as the FEV1 1 hour post-dose of the second bronchodilator minus the FEV1 at 1 hour post-dose of the first bronchodilator. The maximal bronchodilator response for the combination is defined as the FEV1 (the maximal amount of air that can be forcefully exhaled in one second) at 1 hour post-administration of the second bronchodilator minus the corresponding pre-dose FEV1. Derived FEV1 response is FEV1 change from 0 hours (0H) for the first agent assessment (at 1 hour [1H]); change from 1H for the second agent assessment (at 2 hours [2H]); and change from 0H for the combination assessment (at 2H). Data were adjusted for FEV1, smoking status, and center.
Time Frame: up to 10 days
Population: Efficacy Population
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 55
Liters
  First agent, albuterol/salbutamol (A/S) | 0.269 (0.0174)
  First agent, ipratropium | 0.243 (0.0174)
  Second agent, A/S | 0.094 (0.0123)
  Second agent, ipratropium | 0.094 (0.0123)
  A/S followed by ipratropium | 0.363 (0.0200)
  Ipratropium followed by A/S | 0.337 (0.0200)

3. Secondary Outcome: Percentage of Days for Which Participants Achieved a >=12% and 200 Milliliter (mL) Increase From Baseline in FEV1
Description: FEV1 is the maximal amount of air that can be forcefully exhaled in one second. During each study period, pre- and post-bronchodilator spirometry for evaluation of FEV1 was performed at study visits as follows: approximately 1 hour after administration of the first bronchodilator (1 hour), and approximately 1 hour after administration of the second short-acting bronchodilator (2 hours).
Time Frame: up to 35 days
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: percentage of days
Groups:
- Ipratropium Follwed by Albuterol/Salbutamol: All participants randomized to receive a sequence of ipratropium (4 puffs; 20 µg per puff) via an MDI followed by albuterol (4 puffs; 90 µg per puff)/salbutamol (4 puffs; 100 µg per puff) via an MDI in either TP1 or TP2
Arm/Group | Albuterol/Salbutamol Followed by Ipratropium | Ipratropium Follwed by Albuterol/Salbutamol
Number analyzed (Participants) | 55 | 55
percentage of days
  Albuterol/Salbutamol (A/S) alone, 1 hour | 58.4 (38.26) | NA (NA) — Participants in this treatment arm received ipratropium as the first bronchodilator; thus, data were not collected for albuterol/salbutamol (A/S) at this time point.
  A/S followed by ipratropium, 2 hours | 71.7 (35.51) | NA (NA) — Participants in this treatment arm received ipratropium followed by A/S; thus, data were not collected for A/S followed by ipratropium.
  Ipratropium alone, 1 hour | NA (NA) — Participants in this treatment arm received A/S as the first bronchodilator; thus, data were not collected for ipratropium at this time point. | 55.4 (39.34)
  Ipratropium followed by A/S, 2 hours | NA (NA) — Participants in this treatment arm received A/S followed by ipratropium; thus, data were not collected for ipratropium followed by A/S. | 69.1 (36.82)

4. Secondary Outcome: Percentage of Days for Which Participants Achieved a Threshold Increase From Baseline in FEV1 of 100 mL, 200 mL, and 250 mL
Description: as for outcome 3
Time Frame: up to 35 days
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Albuterol/Salbutamol Followed by Ipratropium | Ipratropium Follwed by Albuterol/Salbutamol
Number analyzed (Participants) | 55 | 55
percentage of days
  A/S alone, 1 hour, 100 mL | 81.6 (31.35) | NA (NA) — Participants in this treatment arm received ipratropium as the first bronchodilator; thus, data were not collected for albuterol/salbutamol (A/S) at this time point.
  A/S followed by ipratropium, 2 hours, 100 mL | 85.2 (29.92) | NA (NA) — Participants in this treatment arm received ipratropium followed by A/S; thus, data were not collected for A/S followed by ipratropium.
  Ipratropium alone, 1 hour, 100 mL | NA (NA) — Participants in this treatment arm received A/S as the first bronchodilator; thus, data were not collected for ipratropium at this time point. | 72.9 (38.06)
  Ipratropium followed by A/S, 2 hours, 100 mL | NA (NA) — Participants in this treatment arm received A/S followed by ipratropium; thus, data were not collected for ipratropium followed by A/S. | 81.2 (33.46)
  A/S alone, 1 hour, 200 mL | 59.2 (38.20) | NA (NA) — Participants in this treatment arm received ipratropium as the first bronchodilator; thus, data were not collected for albuterol/salbutamol (A/S) at this time point.
  A/S followed by ipratropium, 2 hours, 200 mL | 72.7 (35.25) | NA (NA) — Participants in this treatment arm received ipratropium followed by A/S; thus, data were not collected for A/S followed by ipratropium.
  Ipratropium alone, 1 hour, 200 mL | NA (NA) — Participants in this treatment arm received A/S as the first bronchodilator; thus, data were not collected for ipratropium at this time point. | 56.0 (39.54)
  Ipratropium followed by A/S, 2 hours, 200 mL | NA (NA) — Participants in this treatment arm received A/S followed by ipratropium; thus, data were not collected for ipratropium followed by A/S. | 70.5 (36.23)
  A/S alone, 1 hour, 250 mL | 45.9 (38.85) | NA (NA) — Participants in this treatment arm received ipratropium as the first bronchodilator; thus, data were not collected for albuterol/salbutamol (A/S) at this time point.
  A/S followed by ipratropium, 2 hours, 250 mL | 64.0 (39.08) | NA (NA) — Participants in this treatment arm received ipratropium followed by A/S; thus, data were not collected for A/S followed by ipratropium.
  Ipratropium alone, 1 hour, 250 mL | NA (NA) — Participants in this treatment arm received A/S as the first bronchodilator; thus, data were not collected for ipratropium at this time point. | 45.8 (36.94)
  Ipratropium followed by A/S, 2 hours, 250 mL | NA (NA) — Participants in this treatment arm received A/S followed by ipratropium; thus, data were not collected for ipratropium followed by A/S. | 59.6 (38.19)

5. Primary Outcome: Variability in Daily FEV1, Estimated by Half Range (i.e., Half the Difference Between Maximum and Minimum Values)
Description: FEV1 is the maximal amount of air that can be forcefully exhaled in one second. During each study period, pre- and post-bronchodilator spirometry for evaluation of FEV1 was performed at study visits as follows: prior to administration of the first short-acting bronchodilator, approximately 1 hour after administration of the first bronchodilator (1 hour), and approximately 1 hour after administration of the second short-acting bronchodilator (2 hours). Variability in daily FEV1 was measured as the fluctuation around the mean FEV1 data collected from Day 1 to Day 10. Variability was measured by the coefficient of variation (CV) and the half range. The CV is the dispersion of the data around the mean, whereas the half range method is half the difference between the maximum and minimum FEV1 values.
Time Frame: up to 10 days
Population: Efficacy Population
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Albuterol/Salbutamol Followed by Ipratropium | Ipratropium Followed by Albuterol/Salbutamol
Number analyzed (Participants) | 55 | 55
Liters
  Pre-dose/non-bronchodilator | 0.136 (0.0627) | 0.135 (0.0780)
  Albuterol/Salbutamol (A/S) alone, 1 hour | 0.125 (0.0525) | NA (NA) — Participants in this treatment arm received ipratropium as the first bronchodilator; thus, data were not collected for albuterol/salbutamol (A/S) at this time point.
  A/S followed by ipratropium, 2 hours | 0.122 (0.0542) | NA (NA) — Participants in this treatment arm received ipratropium followed by A/S; thus, data were not collected for A/S followed by ipratropium.
  Ipratropium alone, 1 hour | NA (NA) — Participants in this treatment arm received A/S as the first bronchodilator; thus, data were not collected for ipratropium at this time point. | 0.145 (0.0805)
  Ipratropium followed by A/S, 2 hours | NA (NA) — Participants in this treatment arm received A/S followed by ipratropium; thus, data were not collected for ipratropium followed by A/S. | 0.137 (0.0726)
Statistical Analysis 1: Comparison: Albuterol/Salbutamol Followed by Ipratropium; Test type: Superiority or Other; Adjusted Mean = 0.058, 95% CI [0.049 to 0.067], Standard Error of Mean 0.0046 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ipratropium Followed by Albuterol/Salbutamol; Test type: Superiority or Other; Adjusted Mean = 0.071, 95% CI [0.062 to 0.080], Standard Error of Mean 0.0046 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Albuterol/Salbutamol Followed by Ipratropium; Test type: Superiority or Other; Adjusted Mean = 0.053, 95% CI [0.044 to 0.062], Standard Error of Mean 0.0046 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Ipratropium Followed by Albuterol/Salbutamol; Test type: Superiority or Other; Adjusted Mean = 0.062, 95% CI [0.053 to 0.071] — [estimate comment as in outcome 1, analysis 4]

6. Secondary Outcome: Variability in Daily Inspiratory Capacity (IC), Estimated by Coefficient of Variation
Description: IC is the the total amount of air that can be drawn into the lungs after normal expiration. During each study period, pre- and post-bronchodilator spirometry for evaluation of IC was performed at study visits as follows: prior to administration of the first short-acting bronchodilator, approximately 1 hour after administration of the first bronchodilator (1 hour), and approximately 1 hour after administration of the second short-acting bronchodilator (2 hours). Variability in daily IC was measured as the fluctuation around the mean IC data collected from Day 1 to Day 10. Variability was measured by the coefficent of variation (CV) and the half range. The CV is the dispersion of the data around the mean, whereas the half range method is the difference between the maximum and minimum IC values.
Time Frame: up to 10 days
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Albuterol/Salbutamol Followed by Ipratropium | Ipratropium Followed by Albuterol/Salbutamol
Number analyzed (Participants) | 55 | 55
Liters
  Pre-dose/non-bronchodilator | 0.078 (0.0305) | 0.083 (0.0374)
  Albuterol/Salbutamol (A/S) alone, 1 hour | 0.069 (0.0310) | NA (NA) — Participants in this treatment arm received ipratropium as the first bronchodilator; thus, data were not collected for albuterol/salbutamol (A/S) at this time point.
  A/S followed by ipratropium (A+I), 2 hours | 0.070 (0.0373) | NA (NA) — Participants in this treatment arm received ipratropium followed by A/S; thus, data were not collected for A/S followed by ipratropium.
  Ipratropium alone, 1 hour | NA (NA) — Participants in this treatment arm received A/S as the first bronchodilator; thus, data were not collected for ipratropium at this time point. | 0.072 (0.0353)
  Ipratropium followed by A/S (I+A), 2 hours | NA (NA) — Participants in this treatment arm received A/S followed by ipratropium; thus, data were not collected for ipratropium followed by A/S. | 0.066 (0.0307)
Statistical Analysis 1: Comparison: Albuterol/Salbutamol Followed by Ipratropium; Test type: Superiority or Other; Adjusted Mean = 0.067, 95% CI [0.058 to 0.076], Standard Error of Mean 0.0045 — Treatment: A/S alone. A mixed model analysis, with period, treatment (A+I, I+A, Albuterol alone, Ipratropium alone), IC Baseline, smoking status at Screening, and center fitted as fixed effects and participant as a random effect was used
Statistical Analysis 2: Comparison: Ipratropium Followed by Albuterol/Salbutamol; Test type: Superiority or Other; Adjusted Mean = 0.070, 95% CI [0.061 to 0.079], Standard Error of Mean 0.0045 — Treatment: ipratropium alone. A mixed model analysis, with period, treatment (A+I, I+A, Albuterol alone, Ipratropium alone), IC Baseline, smoking status at Screening, and center fitted as fixed effects and participant as a random effect was used
Statistical Analysis 3: Comparison: Albuterol/Salbutamol Followed by Ipratropium; Test type: Superiority or Other; Adjusted Mean = 0.069, 95% CI [0.060 to 0.078], Standard Error of Mean 0.0045 — Treatment: A+I. A mixed model analysis, with period, treatment (A+I, I+A, Albuterol alone, Ipratropium alone), IC Baseline, smoking status at Screening, and center fitted as fixed effects and participant as a random effect was used
Statistical Analysis 4: Comparison: Ipratropium Followed by Albuterol/Salbutamol; Test type: Superiority or Other; Adjusted Mean = 0.064, 95% CI [0.055 to 0.073], Standard Error of Mean 0.0045 — Treatment: I+A. A mixed model analysis, with period, treatment (A+I, I+A, Albuterol alone, Ipratropium alone), IC Baseline, smoking status at Screening, and center fitted as fixed effects and participant as a random effect was used

7. Secondary Outcome: Variability in Daily IC, Estimated by Half Range (i.e., Half the Difference Between Maximum and Minimum)
Description: IC is the the total amount of air that can be drawn into the lungs after normal expiration. During each study period, pre- and post-bronchodilator spirometry for evaluation of IC was performed at study visits as follows: prior to administration of the first short-acting bronchodilator, approximately 1 hour after administration of the first bronchodilator (1 hour), and approximately 1 hour after administration of the second short-acting bronchodilator (2 hours). Variability in daily IC was measured as the fluctuation around the mean IC data collected from Day 1 to Day 10. Variability was measured by the coefficent of variation (CV) and the half range. The CV is the dispersion of the data around the mean, whereas the half range method is half the difference between the maximum and minimum IC values.
Time Frame: up to 10 days
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Albuterol/Salbutamol Followed by Ipratropium | Ipratropium Followed by Albuterol/Salbutamol
Number analyzed (Participants) | 55 | 55
Liters
  Pre-dose/non-bronchodilator | 0.225 (0.1017) | 0.236 (0.1166)
  Albuterol/Salbutamol (A/S) alone, 1 hour | 0.229 (0.1004) | NA (NA) — Participants in this treatment arm received ipratropium as the first bronchodilator; thus, data were not collected for albuterol/salbutamol (A/S) at this time point.
  A/S followed by ipratropium, 2 hours | 0.233 (0.1132) | NA (NA) — Participants in this treatment arm received ipratropium followed by A/S; thus, data were not collected for A/S followed by ipratropium.
  Ipratropium alone, 1 hour | NA (NA) — Participants in this treatment arm received A/S as the first bronchodilator; thus, data were not collected for ipratropium at this time point. | 0.235 (0.1026)
  Ipratropium followed by A/S, 2 hours | NA (NA) — Participants in this treatment arm received A/S followed by ipratropium; thus, data were not collected for ipratropium followed by A/S. | 0.221 (0.1066)
Statistical Analysis 1: Comparison: Albuterol/Salbutamol Followed by Ipratropium; Test type: Superiority or Other; Adjusted Mean = 0.228, 95% CI [0.200 to 0.255], Standard Error of Mean 0.0140 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Ipratropium Followed by Albuterol/Salbutamol; Test type: Superiority or Other; Adjusted Mean = 0.231, 95% CI [0.203 to 0.258], Standard Error of Mean 0.0140 — [estimate comment as in outcome 6, analysis 2]
Statistical Analysis 3: Comparison: Albuterol/Salbutamol Followed by Ipratropium; Test type: Superiority or Other; Adjusted Mean = 0.232, 95% CI [0.204 to 0.259], Standard Error of Mean 0.0140 — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 4: Comparison: Ipratropium Followed by Albuterol/Salbutamol; Test type: Superiority or Other; Adjusted Mean = 0.217, 95% CI [0.190 to 0.245], Standard Error of Mean 0.0140 — [estimate comment as in outcome 6, analysis 4]

ADVERSE EVENTS:
Arm/Group | All Randomized Participants
Serious Adverse Events (participants affected / at risk) | 1/56
Other Adverse Events (participants affected / at risk) | 16/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Randomized Participants (N=56)
Death (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Randomized Participants (N=56)
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Bacterial infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.